CLINICAL TRIAL: NCT03033901
Title: Comparison of Sleep Apnea Assessment Strategies to Maximize TBI Rehabilitation Participation and Outcome
Acronym: C-SAS
Status: Completed | Type: Observational
Sponsor: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Craig Hospital (Other); Moss Rehabilitation Research Institute (Other); University of Washington (Other); Baylor Institute for Rehabilitation (Other); Ohio State University (Other); University of South Florida (Other); Palo Alto Veterans Institute for Research (Other); North Florida Foundation for Research and Education (Other)
Responsible Party: Sponsor
Other Study IDs: CER-1511-33005
Record Dates: First submitted 2017-01-18; First posted 2017-01-27 (Estimated); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Apnea, Sleep; Brain Injury, Traumatic
Keywords: Veterans; Comparative Effectiveness Research; Diagnosis
MeSH Terms: conditions — Sleep Apnea Syndromes; Brain Injuries, Traumatic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Polysomnography - Level 1 and Level 3 — Participants will undergo simultaneous administration of Level 1 and 3 polysomnography on the rehabilitation unit with study funded sleep technologist present to meet Level 1 standards.
  Other Names: Philips Respironics Alice 6 Lab Diagnostic System; Nox T3
Device: Actigraphy monitoring — Participants will undergo actigraphy monitoring to assess habitual sleep duration to determine readiness for polysomnography and examine trajectory and duration of sleep.
  Other Names: Philips Respironics Airway (AW) Spectrum Plus Actiwatch
Other: Sleep Apnea Screening — Participants and their family member or proxy, and clinical staff will be asked to answer questions in order to complete the three standardized sleep apnea screening measures.
  Other Names: Berlin Questionnaire; STOPBang Questionnaire; Multivariate Apnea Prediction Index

SUMMARY:
Background: Sleep disorders, including sleep apnea, are common after traumatic brain injury and affect recovery and negatively influence participation in rehabilitation. Sleep apnea is a breathing problem while persons sleep and causes further brain damage and problems with thinking, daily functioning, and overall health. Earlier diagnosis and treatment is important for traumatic brain injury (TBI) survivors to maximize the recovery process. There is little information that guides TBI doctors on how to identify sleep apnea during inpatient TBI rehabilitation, a phase in which people experience the potential for a rapid pace of improvement. The Agency for Healthcare Research has highlighted gaps in best methods for identifying sleep apnea and separately in helping consumers with TBI rehabilitation choices. Partnering with survivors, caregivers, and administrators, investigators developed this study to compare sleep apnea screening and diagnostic tools in TBI rehabilitation settings. This information will provide clinicians, providers, and patients with the best information for early identification of sleep apnea to remove negative influence on the pace of recovery in early phases after TBI.

The Goal: Investigators will compare existing screening (Aim 1) and diagnostic tools (Aim 2) in TBI patients undergoing inpatient rehabilitation. For the second aim, investigators will determine if a more accessible diagnostic test is sufficient to diagnose sleep apnea compared to the traditional method used which is less accessible to consumers. If the more accessible test is good enough, this will increase recognition of this problem and increase patient access to earlier sleep apnea treatment.

Stakeholders and Products. TBI survivors, caregivers, researchers, and policymakers working together on this study helped develop the study questions. Idea exchanges included ways to reach clinicians and TBI survivors/caregivers via existing educational programming and online tools for consumers such as fact sheets and patient/caregiver-focused videos. Other traditional methods will include targeting professional magazines, conferences, and research journals that reach professionals working with TBI survivors and their families at the time of admission to rehabilitation and during the recovery process. This study will occur at rehabilitation hospitals around the country who enroll TBI survivors into a lifetime study called the TBI Model System funded by the Department of Health and Human Services and Veterans Affairs (VA).

DETAILED DESCRIPTION:
Background and Significance:

Meta-analyses of TBI studies found prevalence of obstructive sleep apnea (OSA) was 12 times higher than community-based studies. Yet, sleep apnea in those with TBI is largely undiagnosed. Given that sleep is critical for neural repair and disordered sleep may play a role in slowing functional recovery and prolonging rehabilitation, early detection of sleep apnea is critical (Stakeholder Input). Minimal guidance exists informing TBI and sleep medicine physicians regarding assessment of sleep disorders in the acute rehabilitation setting. The Agency for Healthcare Research and Quality's (AHRQ) Comparative Effectiveness Review highlighted insufficient comparative effectiveness evidence for diagnostic and screening tools. This study proposes to leverage the existing TBI Model System research consortium (TBIMS), funded by the Departments of Health and Human Services and Veterans Affairs, to improve early detection of sleep apnea in patients with TBI undergoing inpatient rehabilitation at six study sites. Study aims are focused around components of phased testing for sleep apnea. Findings will inform clinician's decisions for screening and diagnostic tests to facilitate earlier recognition of sleep apnea (outcome) and subsequently prescribe appropriate treatments.

Study Aims:

Aim I: (Screening) For individuals with TBI, determine comparative effectiveness of 2 American Academy of Sleep Medicine (AASM) endorsed screening tools (STOPBang Questionnaire [STOPBang] vs. Actigraphy [ACG]) to identify those at high risk of sleep apnea as diagnosed through Level 1 polysomnography (PSG). Long-term Objectives: To inform clinician's choices for screening measures to determine presence of sleep apnea.

Exploratory Aim:

Evaluate alternative screening tools (Berlin Questionnaire, Multivariate Apnea Prediction Index [MAPI]) to Level 1 PSG in Aim 1.

Aim II: (Diagnosis) This study will determine the diagnostic accuracy (non-inferiority) of Level 3 PSG in determining presence of sleep apnea in patients with acute TBI patients in the rehabilitation setting. Level 1 PSG will be used as the criterion standard. Long-term Objectives: To inform clinician's choices of diagnostic tests to determine presence of sleep apnea and prescribe appropriate treatments. If Level 3 portable PSG is equivalent to the less accessible Level 1 PSG, this will increase consumer accessibility.

Study Design:

This is a 3-year, multi-center prospective observational cohort study.

Intervention and Comparators:

In Aim I, the screening tools STOPBang and ACG will be compared against one another to determine their sensitivity and specificity in identifying patients with TBI at risk for sleep apnea. In Aim II, the non-inferiority of Level 3 PSG in determining presence and severity of sleep apnea in patients with moderate to severe TBI will be compared to Level 1 PSG.

Study Population:

Consecutive participants to neurorehabilitation at an existing National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR) or VA funded TBIMS Center will make up the study population. Patients will be age 16 and older (18 or older at VA sites), with moderate to severe TBI, admitted for rehabilitation in a U.S. TBIMS inpatient rehabilitation facility, and sleeping > 2 hours/night suggesting habitual sleep duration. Based on historical data from the six study sites participating in this study, investigators in this study conservatively estimated that 70% of patients admitted for inpatient TBI rehabilitation would consent into this study (N=20/month), resulting in a 13-month enrollment estimate of 259 patients. Power analyses of each study aim suggest that a sample size of 237 is the largest sample size needed for sufficient power. The sites participating in this study aim to collectively enroll 259 patients to account for possible further attrition. Based on TBIMS data acquired over the past 25-years, 44% of the sample is female, 64% are categorized as Non-White, median age is 38 years, with predominantly moderate to severe TBI.

Primary outcomes consist of:

1) Positive predictive power of screening tools: STOPBang and ACG, 2) Equivalency in detection of sleep apnea via Level 1 and Level 3 PSG, with diagnosis of sleep apnea based on overall apnea-hypopnea index (AHI) > 5.

Analytic Methods:

Aim 1: Investigators expect that STOPBang values > 5 and abnormal ACG total sleep time (< 5 hours with desaturation) will produce sufficiently high SEs with reasonable tradeoff in SP (noting that SE and SP are inversely related). Similarly, for Level 1 PSG, a diagnosis of sleep apnea will be made if AHI ≥ 5. Cross-tabulations of STOPBang and ACG screening for high risk of sleep apnea (positive/negative) versus Level 1 PSG diagnosis (positive/negative) will be constructed and estimates of diagnostic accuracy (i.e., sensitivity, specificity, positive and negative predictive values, and diagnostic accuracy) will be estimated along with 95% confidence intervals. To address hypothesis 1.1, two-sided McNemar's tests will be used to compare the paired SEs and paired SPs between STOPBang and ACG assuming a significance level of α = 0.05.

Aim 2: The sensitivity (SE) and specificity (SP) of Level 3 PSG (compared to Level 1 PSG, the reference gold standard) will each be estimated and compared to fixed hypothesized rates of SE and SP of 90% and 60%, respectively, considered sufficiently large enough. Level 1 PSG (reference) diagnosis of sleep apnea will be made based on AHI ≥ 5. Level 3 PSG (test) diagnosis will be made based AHI ≥ 5. A cross-tabulation of Level 3 PSG (positive/negative) versus Level 1 PSG (positive/negative) will be constructed and standard measures of diagnostic accuracy will be estimated along with 95% confidence intervals (i.e., sensitivity, specificity, positive and negative predictive values, and diagnostic accuracy).To test for non-inferiority of the SE to 90% and the SP to 60%, a non-inferiority threshold of 0.1 is assumed. If the lower bound on the 95% confidence interval for SE is strictly above 80% and the lower bound on the confidence interval for SP is strictly above 50% then non-inferiority of Level 3 PSG (compared to Level 3 PSG) can be established.

ELIGIBILITY:
Inclusion Criteria:

1. Meet case definition for TBI:

   (A). VA (for James A. Haley Veterans' Hospital): i. Persons fitting the definition of traumatic brain injury (TBI), defined as a traumatically induced structural brain injury, brain trauma, or damage to brain tissue, and/or physiological disruption of brain function as a result of an external mechanical force (also including acceleration/deceleration movement without direct external trauma to the head, a foreign body penetrating the brain, forces generated from events such as a blast or explosion, or other force) as evidenced by self-reported or medically documented (physical examination or mental status examination) new onset or worsening of at least one of the following clinical signs immediately following the event: (a) a period of loss of or a decreased level of consciousness; (b) alteration in mental state at the time of the injury (confusion, disorientation, slowed thinking); (c) loss of memory for events immediately before or after the injury; (d) posttraumatic amnesia (PTA); (d)neurological deficits (weakness, imbalance, change in vision, praxis, paresis/plegia, sensory loss, aphasia, etc.) that may or may not be transient; or (e) intracranial lesion. ii. Age 18 or older at the time of index TBI. iii. Admitted to one of the five designated VA Polytrauma Rehabilitation Centers (PRCs) for comprehensive rehabilitation with the presenting diagnoses of TBI. Comprehensive rehabilitation must occur in the PRC and meet the following criteria: (a) Medical and rehabilitation care are supervised on a regular basis by a physician affiliated with the PRC; (b) 24-hour nursing care is provided to the patient; (c) Physical Therapy (PT), Occupational Therapy (OT), Speech, Rehabilitation Psychology, Neuropsychology, and/or family support/education are provided in an integrated team approach with the expectation of further gain; (d) Operates in a manner consistent with Commission on Accreditation of Rehabilitation Facilities (CARF) standards for brain injury inpatient rehabilitation and/or Medicare requirements for inpatient rehabilitation.

   OR

   (B). Civilian (for civilian sites): Damage to brain tissue caused by an external mechanical force, alteration of consciousness > 24 hours, or loss of consciousness >30 minutes, or Glasgow Coma Scale (GCS) score in the Emergency Department of3-12, or intracranial abnormalities on imaging regardless of GCS;

   AND
2. admission to an inpatient brain injury rehabilitation program;
3. minimum age 16 years at civilian sites and 18 years at the VA site;
4. Understands and provides informed consent to participate (or, if unable, healthcare proxy / legal guardian understands and provides informed consent for the patient);
5. sleep duration > 2 hours/night.

Although not specifically targeted, pregnant women and people with intellectual developmental disorders or prior psychiatric histories meeting the above inclusion/exclusion criteria can be enrolled in this study. Individuals with known history of sleep apnea will be eligible for the study and apnea status will be reconfirmed with new diagnostic study.

Exclusion Criteria:

1. persons less than 16 years old at civilian sites and less than 18 years old at VA site will not be included;
2. pre-injury diagnosis of narcolepsy or persistent daytime somnolence as documented in patient's medical record and/or family report; and/or
3. tracheostomy placed and decannulation or overnight capping of the tracheostomy not feasible during rehabilitation hospitalization.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be TBI patients admitted to inpatient rehabilitation at an existing NIDILRR or VA funded TBI Model System Center who meet study inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Risa Richardson, PhD, Principal Investigator — James A. Haley Veterans' Hospital
Locations (6):
- United States (6):
  - Craig Hospital, Englewood, Colorado
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - The Ohio State University, Columbus, Ohio
  - Albert Einstein Healthcare Network/Moss Rehabilitation Hospital, Elkins Park, Pennsylvania
  - Baylor Institute for Rehabilitation, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Final de-identified data sets underlying publications resulting from the proposed research will be available outside VA in electronic format, through email upon request, after results are published. Data sets will be available for collaborators and other investigators upon request prior to publication (expected time period: 120 days post request). The extent of the data will be de-identified aggregate data only.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available upon request following publication of the primary aims. Data will be made available while the Institutional Review Board (IRB) protocol remains active.
Access Criteria: Data requests will be reviewed by the Study PI and responded to within 120 days of request. Data requests will follow the TBI Model System External Request Standard Operating Procedure (SOP) which is available at www.tbindsc.org.
URL: http://www.tbindsc.org

REFERENCES:
- [Background] Holcomb EM, Schwartz DJ, McCarthy M, Thomas B, Barnett SD, Nakase-Richardson R. Incidence, Characterization, and Predictors of Sleep Apnea in Consecutive Brain Injury Rehabilitation Admissions. J Head Trauma Rehabil. 2016 Mar-Apr;31(2):82-100. doi: 10.1097/HTR.0000000000000230. PMID 26959663
- [Background] Kamper JE, Garofano J, Schwartz DJ, Silva MA, Zeitzer J, Modarres M, Barnett SD, Nakase-Richardson R. Concordance of Actigraphy With Polysomnography in Traumatic Brain Injury Neurorehabilitation Admissions. J Head Trauma Rehabil. 2016 Mar-Apr;31(2):117-25. doi: 10.1097/HTR.0000000000000215. PMID 26959665
- [Background] Towns SJ, Zeitzer J, Kamper J, Holcomb E, Silva MA, Schwartz DJ, Nakase-Richardson R. Implementation of Actigraphy in Acute Traumatic Brain Injury (TBI) Neurorehabilitation Admissions: A Veterans Administration TBI Model Systems Feasibility Study. PM R. 2016 Nov;8(11):1046-1054. doi: 10.1016/j.pmrj.2016.04.005. Epub 2016 May 10. PMID 27178377
- [Background] Nakase-Richardson R. Improving the Significance and Direction of Sleep Management in Traumatic Brain Injury. J Head Trauma Rehabil. 2016 Mar-Apr;31(2):79-81. doi: 10.1097/HTR.0000000000000235. No abstract available. PMID 26959662
- [Background] Holcomb EM, Towns S, Kamper JE, Barnett SD, Sherer M, Evans C, Nakase-Richardson R. The Relationship Between Sleep-Wake Cycle Disturbance and Trajectory of Cognitive Recovery During Acute Traumatic Brain Injury. J Head Trauma Rehabil. 2016 Mar-Apr;31(2):108-16. doi: 10.1097/HTR.0000000000000206. PMID 26709584
- [Background] Nakase-Richardson R, Sherer M, Barnett SD, Yablon SA, Evans CC, Kretzmer T, Schwartz DJ, Modarres M. Prospective evaluation of the nature, course, and impact of acute sleep abnormality after traumatic brain injury. Arch Phys Med Rehabil. 2013 May;94(5):875-82. doi: 10.1016/j.apmr.2013.01.001. Epub 2013 Jan 4. PMID 23296143
- [Background] Silva MA, Nakase-Richardson R, Sherer M, Barnett SD, Evans CC, Yablon SA. Posttraumatic confusion predicts patient cooperation during traumatic brain injury rehabilitation. Am J Phys Med Rehabil. 2012 Oct;91(10):890-3. doi: 10.1097/PHM.0b013e31825a1648. PMID 22660372
- [Background] Nakase-Thompson R, Sherer M, Yablon SA, Nick TG, Trzepacz PT. Acute confusion following traumatic brain injury. Brain Inj. 2004 Feb;18(2):131-42. doi: 10.1080/0269905031000149542. PMID 14660226
- [Background] Nakase-Richardson R, Dahdah MN, Almeida E, Ricketti P, Silva MA, Calero K, Magalang U, Schwartz DJ. Concordance between current American Academy of Sleep Medicine and Centers for Medicare and Medicare scoring criteria for obstructive sleep apnea in hospitalized persons with traumatic brain injury: a VA TBI Model System study. J Clin Sleep Med. 2020 Jun 15;16(6):879-888. doi: 10.5664/jcsm.8352. PMID 32043962
- [Background] Nakase-Richardson R, Schwartz DJ, Ketchum JM, Drasher-Phillips L, Dahdah MN, Monden KR, Bell K, Hoffman J, Whyte J, Bogner J, Calero K, Magalang U. Comparison of Diagnostic Sleep Studies in Hospitalized Neurorehabilitation Patients With Moderate to Severe Traumatic Brain Injury. Chest. 2020 Oct;158(4):1689-1700. doi: 10.1016/j.chest.2020.03.083. Epub 2020 May 6. PMID 32387522
- [Background] Nakase-Richardson R, Hoffman JM, Magalang U, Almeida E, Schwartz DJ, Drasher-Phillips L, Ketchum JM, Whyte J, Bogner J, Dismuke-Greer CE. Cost-Benefit Analysis From the Payor's Perspective for Screening and Diagnosing Obstructive Sleep Apnea During Inpatient Rehabilitation for Moderate to Severe TBI. Arch Phys Med Rehabil. 2020 Sep;101(9):1497-1508. doi: 10.1016/j.apmr.2020.03.020. Epub 2020 May 4. PMID 32376325
- [Background] Zeitzer JM, Hon F, Whyte J, Monden KR, Bogner J, Dahdah M, Wittine L, Bell KR, Nakase-Richardson R. Coherence Between Sleep Detection by Actigraphy and Polysomnography in a Multi-Center, Inpatient Cohort of Individuals with Traumatic Brain Injury. PM R. 2020 Dec;12(12):1205-1213. doi: 10.1002/pmrj.12353. Epub 2020 Mar 26. PMID 32125095
- [Derived] Martin AM, Pinto SM, Tang X, Hoffman JM, Wittine L, Walker WC, Schwartz DJ, Kane G, Takagishi SC, Nakase-Richardson R. Associations between early sleep-disordered breathing following moderate-to-severe traumatic brain injury and long-term chronic pain status: a Traumatic Brain Injury Model Systems study. J Clin Sleep Med. 2023 Jan 1;19(1):135-143. doi: 10.5664/jcsm.10278. PMID 36591795
- [Derived] Steward KA, Silva MA, Maduri P, Tang X, Wittine L, Dams-O'Connor K, Nakase-Richardson R. Obstructive sleep apnea is associated with worse cognitive outcomes in acute moderate-to-severe traumatic brain injury: A TBI Model Systems study. Sleep Med. 2022 Dec;100:454-461. doi: 10.1016/j.sleep.2022.09.012. Epub 2022 Oct 5. PMID 36252414
- [Derived] Martin AM, Almeida EJ, Starosta AJ, Hammond FM, Hoffman JM, Schwartz DJ, Fann JR, Bell KR, Nakase-Richardson R. The Impact of Opioid Medications on Sleep Architecture and Nocturnal Respiration During Acute Recovery From Moderate to Severe Traumatic Brain Injury: A TBI Model Systems Study. J Head Trauma Rehabil. 2021 Sep-Oct 01;36(5):374-387. doi: 10.1097/HTR.0000000000000727. PMID 34489388
- [Derived] Nakase-Richardson R, Schwartz DJ, Drasher-Phillips L, Ketchum JM, Calero K, Dahdah MN, Monden KR, Bell K, Magalang U, Hoffman JM, Whyte J, Bogner J, Zeitzer JM. Comparative Effectiveness of Sleep Apnea Screening Instruments During Inpatient Rehabilitation Following Moderate to Severe TBI. Arch Phys Med Rehabil. 2020 Feb;101(2):283-296. doi: 10.1016/j.apmr.2019.09.019. Epub 2019 Nov 6. PMID 31705855
- See also: NIDILRR-funded TBI Model System website — https://www.tbindsc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group: Potential participants were screened for eligibility. Upon meeting study eligibility requirements, they were asked to consent. Upon consenting, they were screened additional study requirements before undergoing polysomnography.
Period: Overall Study
Arm/Group | Single Group
Started | 345
Completed | 248
Not Completed | 97
Not completed — Ineligible for Polysomnography (PSG) | 59
Not completed — Refused PSG | 23
Not completed — Total Sleep Time < 2 hours | 12
Not completed — Missing Oximetry Data | 3

BASELINE CHARACTERISTICS:
Population: Hospitalized moderate to severe traumatic brain injury participants.
Arm/Group | Single Group
Number analyzed (Participants) | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 203
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participant could identify as more than one race/ethnicity and may be counted in more than one race/ethnicity category.
  Participants
    Hispanic | 33
    White | 184
    Black | 49
    Asian | 8
    Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 248

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index (AHI)
Description: A diagnosis of sleep apnea will be determined by overall apnea-hypopnea index (AHI) greater or equal to 5 and greater than or equal to 15 denoting different severity levels of disease.
Time Frame: During inpatient brain injury rehabilitation, which can occur on average (median) up to 37 days post-traumatic brain injury (TBI) in civilian settings and 132 days in Veterans Affairs (VA) settings.
Measure: Mean (Standard Deviation); unit: times per hour
Arm/Group | Single Group
Number analyzed (Participants) | 248
times per hour | 24.4 (5.4)

2. Other Pre Specified Outcome: STOPBang Sleep Apnea Risk
Description: Sleep apnea screening measure. Risk based on responses to 8 items (2,low risk; 3-4, intermediate risk; >5, high risk).
Time Frame: During inpatient brain injury rehabilitation, which can occur on average (median) up to 37 days post-TBI in civilian settings and 132 days in VA settings.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 248
units on a scale | 2.56 (1.30)

3. Other Pre Specified Outcome: Berlin Sleep Apnea Risk
Description: Sleep apnea screening measure with 10-items. Risk stratification is based on number of items: no risk (no items endorsed), low (endorsement of 1 item) or high risk (endorsement of 2 or more items).
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Single Group
Number analyzed (Participants) | 248
participants
  High risk: 2 categories positive | 54
  Low risk: 1 category positive | 119
  Missing | 75

4. Other Pre Specified Outcome: Actigraphy
Description: Philips brand Actiwatch Spectrum used to measure total sleep time
Time Frame: as for outcome 2
Population: N with complete data = 245. N missing = 3.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Single Group
Number analyzed (Participants) | 245
minutes | 404.7 (74.3)

5. Other Pre Specified Outcome: Multivariate Apnea Prediction Index (MAPI)
Description: The questionnaire consists of 3 breathing-related questions and information on demographics (sex, weight, height, age), from which a probability of having sleep apnea (0%-100%) can be calculated. The test-retest reliability of the breathing questions is 0.92 and has a good internal consistency with Cronbach a of 0.85-0.93. A MAPI score of 0.50 (ie, calculated 0% likelihood of having clinically significant sleep apnea with a Respiratory Distress Index>10) has a 0.88 sensitivity and 0.55 specificity.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent probability
Arm/Group | Single Group
Number analyzed (Participants) | 248
percent probability | 0.23 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse events time frame was between May 1, 2017 (starting enrollment) until February 1, 2020 (end of study). For each participant, adverse events monitoring occurred between time of study enrollment and either (1) time completed all study procedures, or (2) time participant withdrew from study. The adverse event monitoring period lasted for 2 years and 9 months. For the study sample as a whole, the average monitoring period was 8 days.
Description: The definitions used during the study match the clinicaltrials.gov definitions.
Arm/Group | Single Group
All-Cause Mortality (participants affected / at risk) | 0/248
Serious Adverse Events (participants affected / at risk) | 0/248
Other Adverse Events (participants affected / at risk) | 0/248

LIMITATIONS AND CAVEATS:
The sample may not represent the full population of inpatient rehabilitation patients with TBI; Short lengths of stay impacted study participation; unclear if findings extend to chronic phases of TBI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT03033901/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT03033901/SAP_001.pdf